CLINICAL TRIAL: NCT02916459
Title: Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA) Versus Flexible 19G Endobronchial Ultrasound Transbronchial Needle (Flex 19G EBUS-TBNA) in the Assessment of Mediastinal and Hilar Lymph-adenopathy: a Randomised Trial
Brief Title: EBUS-TBNA vs Flex 19G EBUS-TBNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Principal Investigator, Felix JF Herth, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 19G 1.1-2016
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Lymphadenopathy; Lung Cancer; Sarcoidosis; Lymphoma
MeSH Terms: conditions — Lymphadenopathy; Lung Neoplasms; Sarcoidosis; Lymphoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- EBUS-TBNA (Active Comparator): Mediastinal and hilar lymph node sampling using a standard 21G EBUS-TBNA needle
  Interventions: Device: 21G EBUS-TBNA needle
- Flex 19G EBUS-TBNA (Experimental): Mediastinal and hilar lymph node sampling using the flexible 19G EBUS-TBNA needle
  Interventions: Device: Flexible 19G EBUS-TBNA needle

INTERVENTIONS:
Device: 21G EBUS-TBNA needle
  Arms: EBUS-TBNA
Device: Flexible 19G EBUS-TBNA needle
  Arms: Flex 19G EBUS-TBNA

SUMMARY:
This is a prospective randomised diagnostic clinical study to determine whether the use of a new flexible sampling needle can improve the yield of endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA). Patients undergoing EBUS-TBNA for clinical reasons as deemed necessary by the managing physician or multidisciplinary team will be randomised to undergo either EBUS-TBNA or Flex 19G EBUS-TBNA. The procedure will be performed under local anaesthesia using conscious sedation or general anaesthesia according to usual practice at the trial centre. Specimens will be placed in saline and formalin and forwarded to the pathology laboratory. The specimens will be spun down to create a cell pellet which will undergo cytological and histological examination as per usual protocol at the trial centre.The pathologist, who will be blinded as to which technique was used to obtain the sample, will grade the quality, quantity, and cellularity of the specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for EBUS-TBNA as part of clinical care
2. Lymph nodes larger than 10mm in diameter
3. Age > 18 years
4. written informed consent

Exclusion Criteria:

1. Contraindication to needle biopsy (e.g. coagulopathy, anticoagulation, thrombocytopenia)
2. Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The difference in quality of diagnostic tissue obtained between the two study arms following 4 separate needle punctures per lymph node | 1 week
  Both specimens (cell pellet and tissue fragments) will be assessed by means of a semiquantitative assessment of material (normal lymph node or lesional tissue) present using the formal scoring system described by Mair

SECONDARY OUTCOMES:
The difference between the two study arms in the percentage of lymph nodes sampled where enough tissue is obtained for complete immunohistochemical and genetic mutation analysis | 1 week
The difference in complication rates between the two study arms | 1 month
The difference between the two study arms in yield (quantity of diagnostic material) in patients ultimately diagnosed with sarcoidosis | 1 week
The difference between the two study arms in yield (quantity of diagnostic material) in patients ultimately diagnosed with lymphoma | 1 week
The difference in sensitivity for detecting sarcoidosis between the two study arms | 1 week
  Sensitivity = True Positives/(True Positives + False Negatives)
The difference in sensitivity for detecting lymphoma between the two study arms | 1 week
  Sensitivity = True Positives/(True Positives + False Negatives)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pneumology and Critical Care medicine, Heidelberg, Baden-Wurttemberg, Germany